CLINICAL TRIAL: NCT04027322
Title: Inhaled Glucocorticoids for Acute Pharyngitis: A Randomized Clinical Trial
Brief Title: Inhaled Steroids for Acute Pharyngitis.
Acronym: ISAP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Oman Medical Speciality Board (Other Government)
Responsible Party: Principal Investigator, Al Yaqdhan Al Atbi, Emergency Medicine Specialist, Royal Oman Police Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OMSB
Record Dates: First submitted 2019-07-18; First posted 2019-07-19 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Acute Pharyngitis
Keywords: Pharyngitis; Sore Throat; Glucocorticoids; Nebulizers
MeSH Terms: conditions — Pharyngitis | interventions — Budesonide; Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Budesonide (Active Comparator): Drug Name: budesonide Dose: 2000mcg (2mg) of budesonide nebulizer solution is mixed with normal saline solution to make a total volume of 8mL.
  Frequency: Stat Dose Route: Nebulization
  Interventions: Drug: Budesonide 0.25 MG/ML Inhalant Solution
- Dexamethasone (Active Comparator): Drug Name: Dexamethasone Sodium phosphate Dose: 8mg of IV formula of dexamethasone is mixed with normal saline to make a total volume of 8ml.
  Frequency: Stat Dose Route: Nebulization
  Interventions: Drug: Dexamethasone
- Control (Placebo Comparator): Drug Name: Normal Saline Dose: 8ml. Frequency: Stat Dose Route: Nebulization
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Budesonide 0.25 MG/ML Inhalant Solution — Both medications used for the intervention groups are Glucocorticoids. The effect of glucocorticoids in AP can be attributed to their anti-inflammatory actions. They inhabit the formation of the pro-inflammatory mediators in the endothelial cells of the airways. This will decreases the inflammatory reaction at the pharynges which result in a reduction of throat pain.
  Studies have shown that the use of a single dose of systemic glucocorticoids for acute pharyngitis did not result in significant adverse events and no serious adverse events were reported (7) (8).
  Arms: Budesonide
Drug: Dexamethasone — Both medications used for the intervention groups are Glucocorticoids. The effect of glucocorticoids in AP can be attributed to their anti-inflammatory actions. They inhabit the formation of the pro-inflammatory mediators in the endothelial cells of the airways. This will decreases the inflammatory reaction at the pharynges which result in a reduction of throat pain.
  Studies have shown that the use of a single dose of systemic glucocorticoids for acute pharyngitis did not result in significant adverse events and no serious adverse events were reported (7) (8).
  Arms: Dexamethasone
Drug: Normal saline — Placebo for the control group.
  Arms: Control

SUMMARY:
Background: Acute pharyngitis (AP) is a common presentation to the Emergency Department (ED). Most AP patients' who present to the ED are interested in relief their sore throat (pain). There are different approaches available in the literature to control AP pain. Studies have shown that the use of systemic glucocorticoids significantly decreases patients' sore throat. Up to our knowledge, there are no available trials looking at the role of nebulized glucocorticoids in treating infective AP.

Aim: Our aim is to investigate in pediatrics and adults population ≥5 years presenting to ED with AP if the use of a single dose of nebulized glucocorticoids as an adjunct to standard AP treatment, compared with placebo leads to complete resolution or improvement in symptoms.

Method: The investigators are planning to conduct a multi-center, double-blind randomized control trial. There will be three arms; first arm: nebulized Budesonide, second arm: nebulized Dexamethasone and third arm: placebo nebulized Normal Saline (NS). The patients will be followed up for 7 days through phone calls to assess the primary and secondary outcomes. Our primary objective is to investigate whether the use of a single dose of nebulized glucocorticoids compared with placebo leads to significant improvement or complete resolution of the sore throat within 24hrs. Our secondary objectives are to assess if a single dose of glucocorticoids will: reduce sore throat at 48 hours, reduce absence from work or school, reduce the incidence of hospital admission, and reduce the rate of re-attendance to ED. Since there is no available data about the effect of nebulized glucocorticoids in AP, the appropriate sample size will be calculated after running a pilot study. The data will be recorded in the EpiData@ software. Then the data will be analyzed using the SPSS@ software. The ethical approval was sought from the ethical committee in each participating hospital and they approved it.

Results: The result of this study will be presented in local conferences as well in international conferences. The investigators will aim to publish the study in a well-known international emergency medicine journal.

Clinical application: up to our knowledge this study is the first study worldwide looking at the effect of nebulized glucocorticoids in patients with infective acute pharyngitis. As mentioned earlier that there are multiple approaches available in the literature to control sore throat pain and if our hypothesis turned to be correct then another alternative treatment can be added. The investigators believe that the use of topical route to administer glucocorticoids is more convenient for physicians and have less chance to develop adverse effect in comparison to systemic steroids.

DETAILED DESCRIPTION:
Introduction:

Acute pharyngitis (AP) is a commonly diagnosed condition in the Emergency Departments (ED). In the United States (USA), there are approximately 12 million visits to health institutions due to acute pharyngitis(1). It is defined as an acute inflammation of the pharynx and/or tonsils and the diagnosis is made clinically(2). Although there are variable etiologies for AP, viral infections are the commonest(3). Symptoms of AP vary in the severity but the most common symptom for which the patients seek medical care is a sore throat. The patient may complain of fever, flu symptoms, odynophagia (painful swallowing), neck pain, poor oral intake, nausea, and vomiting. Of these symptoms, around 80% of patients with AP were interested more to relieve their pain(4).

Different approaches were suggested to control AP pain. It is well established that oral acetaminophen and ibuprofen are effective in decreasing AP pain(5). Different forms of topical therapies like lozenges/drops, throat sprays, gargles, and teas are also available for relief AP related pain. There is no evidence that a particular topical lozenge or spray is superior in efficacy(6).

Systemic glucocorticoids have been proven to be effective in decreasing AP sore throat. Systemic reviews and meta-analysis studies showed that a single dose of systemic glucocorticoids decreases pain within 24 hours by two times and at 48 hours by 1.5 times(7) (8) compared to patients who didn't receive steroids. A recently published trial showed that the use of systemic glucocorticoids in less severe acute pharyngitis significantly result in complete resolution of a sore throat at 48hours(9).

Glucocorticoids are commonly used medication in the emergency department. They have a very good safety profile(10). A short course of glucocorticoids is less likely to result in adverse events (AE) and if occurred usually with systemic, not with local glucocorticoids(10). Studies have shown that the use of a single dose of systemic glucocorticoids for acute pharyngitis did not result in significant adverse events and no serious adverse events were reported (7) (8).

The effect of glucocorticoids in AP can be attributed to their anti-inflammatory actions. They inhabit the formation of the pro-inflammatory mediators in the endothelial cells of the airways. This will decreases the inflammatory reaction at the pharynges which will lead to a reduction in the throat pain.

Up to our knowledge, no available trials are looking at the role of nebulized glucocorticoids in treating infective AP. A Randomized Control Trial (RCT) showed that the use of nebulized dexamethasone significantly decreases the incidence and severity of postoperative sore throat at 2, 4, 8, and12 hours(11). There was no complication reported from the use of nebulized dexamethasone(11). Despite the available evidence about the effectiveness of glucocorticoids in acute pharyngitis, some physicians are still reluctant to prescribe it as an adjunct therapy.

The investigators hypothesized that the uses of local glucocorticoids (nebulization) will significantly reduce sore throat in patients with AP. The investigators believe that the use of topical route to administer glucocorticoids is more convenient for physicians and have less chance to develop adverse effect in comparison to systemic steroids. The investigators aim to investigate in pediatrics and adults population ≥5 years presenting to ED with AP if the use of a single dose of nebulized glucocorticoids as an adjunct to standard AP treatment, compared with placebo leads to complete resolution or improvement in symptoms.

Objectives:

* Primary Objective:

  - To investigate in pediatrics and adults population ≥5 years presenting to ED with AP if the use of a single dose of nebulized glucocorticoids as an adjunct to standard AP treatment compared with placebo leads to significant improvement or complete resolution of the sore throat within 24hrs.
* Secondary objectives:

To investigate whether a single dose of inhaled Glucocorticoids compared with Placebo will:

* Reduce sore throat at 48 hours.
* Reduce absence from work or school.
* Reduce the incidence of hospital admission due to the complication of the sore throat within 7 days.
* Reduce the rate of re-attendance to ED.

Methodology

* Study Design: The trial will be multi-center, double-blind randomized control trial. There will be three arms; first arm: nebulized Budesonide, second arm: nebulized Dexamethasone and third arm: placebo nebulized Normal Saline (NS). The patients will be followed up for 7 days through phone calls to assess the primary and secondary outcomes.

* Target population:

  * Overall Description of Trial Participants:

    * Pediatrics and adult aged 5 years or over presenting to the emergency department (ED) with acute pharyngitis (AP).
  * Inclusion Criteria and Exclusion criteria:

refer to "Eligibility" section.

> The Number of Participants: Up to our knowledge the available literature only about the use of systemic glucocorticoids in AP. No available studies looked at the effect of nebulized glucocorticoids in AP sore throat. Therefore The investigators are conducting a pilot study to look at the effect of nebulized glucocorticoids and from the result of the pilot study, the sample size will be calculated.

The recruitment for the pilot study is already started since June 2019. It is conducted in two centers for 20 participants in each arm. The investigators will use the same protocol (mentioned below) for both the pilot study and the main study.

*Study Procedures:

> Inform consent: After checking for eligibility and patient willingness to participate in the trial, a written informed consent form will be given to the participant by the enrolling clinician. The written informed consent will be submitted to the patient so he/she can read it plus a verbal presentation of the form will be conducted by the care provider. The form has to be signed by the participant or caregiver personally.

Details about the exact nature of the trial, the implications of the trial and possible adverse effects will be included in both verbal presentations and written informed consent. The written consent will clearly state that the participant has the rights to withdraw from the study at any time for any reason without prejudice to future care.

> Screening and Eligibility Assessment: Any patient who presented to the emergency department with a sore throat should be screened by the triage nurse or doctor for eligibility of the participant for the study. A participant information sheet will be kept in the triage room and the doctors' room. The treating physician will check the eligibility of the patient by checking inclusion and exclusion criteria. Any patient who is not eligible to participate or declines to participate will be recorded on the screening log with reasons for ineligibility or declining (if known) and have no further involvement in the trial.

All patients who are found eligible and accept to participate in the trial will be included in the trial and proceed to baseline trial assessment.

* Baseline Trial Assessment:

  * Once the participant is eligible for the trial, the treating physician will take the baseline characteristics.
  * The treating physician will explain to the participant the process of the trial and the ways of data recording. He/she will explain to the participant how to fill the trial dairy which will be provided to them.
  * The treating physician will take the contact number of the participant and inform him/her that he/she will be called by the trial investigators at the following time:
  * At 24 hours, on day 2, and on day 7 after inclusion in the trial.
  * May also receive 1 or 2 calls to encourage the patient to complete the trial and to check on participant's compliance to study protocol.
  * Data collection sheet will be available online using "Google Forms". The treating physician is required to fill the baseline assessment sheet within 6 hours from participant inclusion in the trial and send it through online to the principal investigator.
  * Items to be collected in the baseline data collection sheet:

    * Socio-demographic factors:

      o Age
      * Gander
      * Smoking
    * Medications:

      o Need for antibiotics

      o Any other advised treatment, including Paracetamol, ibuprofen, Gargle, Zinc, steam, and others.
    * Symptoms will include:

      o Duration of sore throat and odynophagia

      o Presence or absence of cough, hoarse voice, coryza, fever in the last 24 hours
    * Clinical examination findings will include:

      o Presence of pharyngeal inflammation

      o Presence of inflamed tonsils without follicles

      o Presence of inflamed tonsils with purulent follicles

      o Presence of tender cervical lymphadenopathy
      * Temperature and type of thermometer used for measuring
    * Throat swab for microscopy and culture: to be collected in the day of presentation.
    * Patient completed items will include:

      * Ratings of throat soreness, pain on swallowing and difficulty swallowing using Numeric pain score.
* Randomization:

  - Sealed non-transparent envelopes with blocked randomization (3,6,9).

  - Envelops contain a folded paper written on it the type of intervention: as follow (Dexamethasone, Budesonide, or Placebo).
  * Each time the care provider decided to include a patient in the study he/she picks an envelope according to the sequence of randomization and read the content of it.
* Blinding:

  * Both the follow-up investigators (the assessors) and the patients will be blinded, but not the treating physician.
  * Method: all patients will receive nebulization of 8 milliliters (ml) solution:

Placebo normal saline will be administered for the control group: dose 8 ml of normal saline.

Glucocorticoid nebulization for the intervention group: Dose of 8 ml of study medications

* After the treating physician includes a patient to the trial, he/she will send the patient's data to the principal investigator through online Google Forms. The principal investigators will assign another investigator to contact the patient without telling him the type of intervention the patient received and ask him/her about the study endpoint outcomes (mentioned above). The study outcome assessors will be required to fill the data online using Google Forms and forward it back to the study principal investigator.

  > Subsequent assessments:
* 3 new phone numbers will be opened for the trials.
* Each participant will be provided with a diary which is specifically designed for the trial. It will include patient questions about patient pain and other symptoms. The patient will keep recording in the diary for 7 days.
* The participants will be contacted by telephone at 24hours, 48hours, and 7 days to collect the study primary and secondary objectives and to ensure completion of symptoms diary.
* The follow-up call is standardized with pre-specified questions
* An additional phone call will be done if needed to encourage the participants to complete symptoms diary.

Definition of End of Trial

- The trial ends once the targeted sample size achieved and follow up completed.

Discontinuation/ Withdrawal of Participants from Study Treatment:

* Each participant has the right to withdraw from the study at any time for any reason.
* The investigators may discontinue a participant from the study for any of the following reasons:

  1. Failure of the participant to follow the study protocol, major missing data e.g. reporting the primary endpoint of the study.
  2. Continuation of the study will harm the patient
* The reason for withdrawing/discontinuation from the study will be recorded in the case report form.
* If the reason for the participant withdraw is an adverse event from the study intervention, a follow-up appointment will be arranged for the participant with study investigators.
* If the participant found to be not eligible for the trial after randomization, he/she will be removed from the trial and all his information will be removed from the trial database.

  * Description of Study Treatment: refer to "Arms and Interventions" section

  * Compliance with Study Treatment:
* The participant will be observed taking the single dose of study medication once they have provided full informed consent.

  * Availability of the Study Treatment:
* The study medications will be supplied by the participating hospitals.
* The study medications are available in the participating hospitals.

  * Concomitant Medication:
* The treating physician may prescribe any of the following medications:

  1. Antibiotics, if indicated
  2. Any other advised treatment, including Paracetamol aspirin ibuprofen, Gargle, Difflam, Zinc, steam, and others.

     * Post-Trial Treatment:
* After study medication administration in ED, the participants follow normal medical care of AP.

  *Safety reporting:
* Glucocorticoids are used Commonly in the emergency department. They have a very good safety profile(10). A short course of glucocorticoids is less likely to result in adverse events and if occurred usually with systemic, not with local glucocorticoids (10). Studies have shown that the use of a single dose of systemic glucocorticoids for acute pharyngitis did not result in significant adverse events and no serious adverse events were reported (7) (8).
* Although the risk of developing adverse events secondary to the usage of nebulized glucocorticoids, all adverse events will be documented by the study investigators. Any adverse events reported by the participant will be investigated for causality. These investigations will be done by a medically qualified investigator. The severity of events will be assessed on the following scale: 1=mild, 2=moderate, 3=severe.
* A participant has the free rights to withdraw from the trial due to what he or she perceives as intolerable adverse events. Adverse events that result in a participant's withdrawal from the study will be recorded on the withdrawal form.

Statistics:

- The data will be recorded in the EpiData@ software. Then the data will be analyzed using the SPSS@ software. All randomized participants will be included in the analysis, assuming no complete resolution for missing data. The proportion of complete resolution of a sore throat at 24 hours in those participants who have received nebulized glucocorticoids on which this trial is powered will be compared using logistic regression model. Odds ratio and their 95% confidence interval (CI) will be reported. The p-value of <0.05 will be considered statistically significant.

Criteria for the Termination of the Trial:

The trial will be terminated in case of the following:

- If the study medications appear to be harmful to the participants e.g. multiple cases reported serious adverse events

Quality Control and Quality Assurance Procedures:

- The study will be conducted according to this protocol. All the investigators will receive training on the trial procedure before the start. The principal investigator will be responsible for continuous monitoring of compliance with the study protocol and data recording.

Ethics:

* The study will be conducted in three hospitals in Muscat. Two hospitals are under the umbrella of Armed Forced Hospital (AFH) and one hospital is the Royal Oman Police Hospital (ROP). The ethical approval was sought from each hospital individually and they approved it.
* Trial staff will ensure that the participants' anonymity is maintained. Participants' details will be identified by their hospital Identification (ID) number e.g. (AFH_ID number). All data will be stored securely and only accessible by the trial staff.

Finance:

* To conduct such a study, sponsors who will help us to cover the costs of the study is needed. The investigators submitted the proposal to the following institution looking for financial support: The Research Council Oman: status pending
* The investigators asked the participating hospitals for their permission to utilize their resources to conduct the study. The investigators got all the study's medications and equipment from the participating hospitals.

Result dissemination:

- The result of this study will be presented in local conferences as well in international conferences. The investigators will aim to publish the study in a well-known international emergency medicine journal.

ELIGIBILITY:
Inclusion Criteria:

* Pediatrics and adult > 5 years of age
* Patients complain of acute sore throat likely due to infective pharyngitis/tonsillitis as judged by the treating clinician.
* Onset of symptoms within 7 days
* Patient or caregiver has the capacity and willingness to give consent and complete the trial paperwork, including the symptom diary.
* Not on antibiotics for AP.

Exclusion Criteria:

* Pregnant or lactating mother.
* Recent use of oral or inhaled steroids within 7 days.
* Presence of an alternative diagnosis e.g. pneumonia, croup, bronchiolitis,
* Known immune-deficiency (e.g. HIV, active chemotherapy or advanced cancer)
* Complicated acute sore throat that hospital admission is required (e.g. completely unable to swallow, very systemically unwell, or peritonsillar abscess)
* Presence of clear contraindication for steroids use (refer to the British National Formulary (BNF) list of contraindications)
* Requirement for the live vaccine in the next 7 days.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with the complete resolution of sore throat after 24hours from intervention. | 24 hours after intervention.
  Direct report by the patient of presence or absence of complete resolution of sore throat at 24 hours by telephone.

SECONDARY OUTCOMES:
Number of participants with the complete resolution of sore throat after 48 hours from intervention. | 48 hours after intervention.
  Direct report of complete resolution of sore throat at 48 hours.
Number of hours needed until the onset of pain relief. | 7 days after intervention.
  Direct report of time to onset of pain relief in hours within 7 days.
Number of hours needed until complete resolution of sore throat. | 7 days after intervention.
  Direct report of time to complete symptom resolution in hours within 7 days.
Average number of days of absences from work among participants. | 7 days after intervention.
  Time missed from work or education over subsequent 7 days.
Number of participants reattended the Emergeancy Department (ED) due to acute pharyngitis. | 7 days after intervention.
  Attendance at ED within 7 days with symptoms or complications associated with sore throat e.g. peritonsillar abscess
Number of participants developed complications related to acute pharyngitis. | 7 days after intervention.
  Hospital admission with related complications of sore throat within 7 day.

CONTACTS AND LOCATIONS:
Overall Officials: Al Yaqdhan H Al Atbi, EM Resident. PGY 5, Principal Investigator — Oman Medical Board Specialty (OMSB)
Locations (3):
- Oman (3):
  - Armed Forces Hospital, Muscat
  - Mortaafah Armed Medical Hospital (MAM), Muscat
  - Royal Oman Police Hospital, Muscat

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schappert SM, Rechtsteiner EA. Ambulatory medical care utilization estimates for 2006. Natl Health Stat Report. 2008 Aug 6;(8):1-29. PMID 18958997
- [Result] van Driel ML, De Sutter A, Deveugele M, Peersman W, Butler CC, De Meyere M, De Maeseneer J, Christiaens T. Are sore throat patients who hope for antibiotics actually asking for pain relief? Ann Fam Med. 2006 Nov-Dec;4(6):494-9. doi: 10.1370/afm.609. PMID 17148626
- [Result] Schachtel BP, Fillingim JM, Thoden WR, Lane AC, Baybutt RI. Sore throat pain in the evaluation of mild analgesics. Clin Pharmacol Ther. 1988 Dec;44(6):704-11. doi: 10.1038/clpt.1988.215. PMID 3197368
- [Result] Sadeghirad B, Siemieniuk RAC, Brignardello-Petersen R, Papola D, Lytvyn L, Vandvik PO, Merglen A, Guyatt GH, Agoritsas T. Corticosteroids for treatment of sore throat: systematic review and meta-analysis of randomised trials. BMJ. 2017 Sep 20;358:j3887. doi: 10.1136/bmj.j3887. PMID 28931508
- [Result] Hayward G, Thompson MJ, Perera R, Glasziou PP, Del Mar CB, Heneghan CJ. Corticosteroids as standalone or add-on treatment for sore throat. Cochrane Database Syst Rev. 2012 Oct 17;10:CD008268. doi: 10.1002/14651858.CD008268.pub2. PMID 23076943
- [Result] Hayward GN, Hay AD, Moore MV, Jawad S, Williams N, Voysey M, Cook J, Allen J, Thompson M, Little P, Perera R, Wolstenholme J, Harman K, Heneghan C. Effect of Oral Dexamethasone Without Immediate Antibiotics vs Placebo on Acute Sore Throat in Adults: A Randomized Clinical Trial. JAMA. 2017 Apr 18;317(15):1535-1543. doi: 10.1001/jama.2017.3417. PMID 28418482
- [Result] Atef K Salama, Ahmed M El-badawy. Does nebulized dexamethasone decrease the incidence of postextubation sore throat?: a randomized controlled study. Ains Shams J Anesthiology 9(1):104-7, 2016.
- [Result] Fitzgerald D, Mellis C, Johnson M, Allen H, Cooper P, Van Asperen P. Nebulized budesonide is as effective as nebulized adrenaline in moderately severe croup. Pediatrics. 1996 May;97(5):722-5. PMID 8628614
- [Result] Klassen TP, Feldman ME, Watters LK, Sutcliffe T, Rowe PC. Nebulized budesonide for children with mild-to-moderate croup. N Engl J Med. 1994 Aug 4;331(5):285-9. doi: 10.1056/NEJM199408043310501. PMID 8022437
- [Derived] Al Atbi AY, Al Khalasi U, Al Atbi A, Al Rawahi S, Al Shaffi K, Al-Mamari S, Al Sakiti M, Al Mujani S, Al Reesi A, Al Shamsi M. Efficacy of nebulized glucocorticoids for acute pharyngitis in an emergency department outpatient population: a multicenter, double-blind, randomized clinical trial. CJEM. 2025 Jul;27(7):543-550. doi: 10.1007/s43678-025-00906-5. Epub 2025 Apr 24. PMID 40272745
- See also: Wendy Stead. Symptomatic treatment of acute pharyngitis in adults. UPTODATE. 2018 [cited 2019 Jan 7]. — http://www.uptodate.com/contents/symptomatic-treatment-of-acute-pharyngitis-in-adults?search=acute%20pharyngitis&source=search_result&selectedTitle=2~150&usage_type=default&display_rank=2